CLINICAL TRIAL: NCT04020029
Title: Leveraging Mindsets to Improve Health and Wellbeing in Cancer Patients
Brief Title: Leveraging Mindsets to Improve Health and Wellbeing in Patients With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never run due to Covid
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alia Crum, Associate Professor of Psychology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-43605; NCI-2020-00541 (Other: National Cancer Institute: Clinical Trials Reporting Program); NCT03910283 (obsolete NCT alias)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Stress Mindset Measure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindset Intervention (Experimental): Mindset Intervention will include watching three brief ~10-25 minute films and respond to a number of short reflection activities after viewing the films.
  Interventions: Other: Mindset; Other: Reflection activities
- Treatment As Usual (TAU) (Active Comparator): TAU Control Arm will complete the same assessments as those participants in the Mindset Intervention Arm, but will not view the short films or complete the corresponding response activities.
  Interventions: Other: Reflection activities

INTERVENTIONS:
Other: Mindset — Mindset Intervention will include watching three brief ~10-25 minute films
  Arms: Mindset Intervention
Other: Reflection activities — Reflection activity include exercises to internalize the message

SUMMARY:
Primary Objectives:

Mindsets have been rigorously studied in the domains of development, education, and more recently, in health and disease. However, there are no large-scale longitudinal studies of the mindsets held by cancer patients and how they may affect treatment outcomes, physical health, and psychological well-being. This randomized, single-blind, treatment-as-usual (TAU) control study aims to assess (1) mindsets at four time points spanning from the point of diagnosis to six weeks post-treatment to patients who are newly diagnosed with cancer and undergoing treatment with curative intent, and (2) the impact of a brief but targeted mindset intervention to help instill more useful mindsets about the nature of cancer and the role of the body on patient reported measures of physical and psychological health. This study aims to add to the existing literature on psychosocial interventions for cancer patients and survivors while addressing the substantial time and cost limitations of traditional interventions. It also contributes to the body of research indicating that mindsets play an important role in both health and wellbeing.

Secondary Objectives:

This study has two secondary objectives. First, we aim to determine the impact of patient mindsets on measures of treatment (treatment efficacy and treatment related adverse events) and psychosocial health (stress, coping, mood, emotions). Second, we aim to understand the relationship between patient mindsets and biomarkers of immune and inflammatory processes in patients undergoing cancer treatment

ELIGIBILITY:
Inclusion Criteria:

* We will only recruit patients ≥ 18 years who are fluent in English and are without cognitive impairment. We have no gender, race, or ethnicity restrictions. Diagnosis of cancer (breast, lung, GI or colorectal, or lymphoma) and treatment given with curative intent.
* Patients diagnosed with lung cancer, breast cancer, GI/Colorectal cancer, or Lymphoma to be treated with curative intent will be eligible for this study.
* Participants will be recruited if they are receiving at least one course of systemic treatment. As we are recruiting participants near the point of diagnosis, we will target individuals who have not received prior therapy for cancer.
* Neither ECOG or Karnofsky Performance Status will be employed
* Ability to understand and willingness to sign a written informed consent document is required for participation in this study.
* Treatment plan includes course of systemic treatment involving no less than 4 and no more than 12 infusions.

Exclusion Criteria:

* Surgical procedures, if applicable, must take place either before the initiation of systemic treatment or after the last infusion.
* There are no restrictions regarding the use of other investigational agents; however, use of any investigational agents will be recorded.
* No active major mental health diagnoses including severe depression, severe anxiety, bipolar / manic depressive disorder, post-traumatic stress disorder, schizophrenia, or any psychotic disorder. Patients with mild depression or anxiety, or depression or anxiety that is well managed with treatment, will not be excluded
* Pregnant / nursing patients will not be excluded from the study
* Patients with a previous diagnosis of cancer (cancer survivors) will be excluded from this study. Cancer survivors may already have preconceived notions about the nature of a cancer diagnosis and the course of treatment, and therefore may not respond to our intervention in the same way as individuals who are encountering a cancer diagnosis for the first time.
* Patients who are HIV-positive will not be excluded.
* Patients who have major comorbidities that would substantially reduce life expectancy despite successful cancer treatment (i.e., comorbid end stage heart disease or kidney disease) will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Survey | 6 weeks
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy (FACT-G), a widely used patient reported health outcome measure. The FACT-G consists of 27 questions. Each question is answered on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Higher scores on the FACT-G indicate better quality of life. Questions fall into four subscales measuring four domains of quality of life: physical wellbeing (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), and functional well-being (7-questions).

SECONDARY OUTCOMES:
Measuring mindsets | 6 weeks
  Patient mindsets will be measured using the Illness Mindset Inventory (IMI). The IMI is a 20-item measure of mindsets about chronic illness. The Cancer version of the IMI consists of two subscales: mindsets about the nature of cancer and mindsets about the role of the body. Each item is rated on a 6 point Likert scale ranging from strongly disagree (1) to strongly agree (6).
Fear of Cancer Recurrence | 6 weeks
  Fear of Cancer Recurrence will be measured using the Cancer Worry Scale (CWS). The CWS is a 6-item measure that assesses worry about the risk of developing cancer in cancer survivors. All items use a 4-point scale of frequency, ranging from 1 (not at all) to 4 (almost all the time). The CWS will be measured at only one time-point (CP-7), 6 weeks after the completion of treatment
Biomarker Analyses | 6 weeks
  Blood samples will be analyzed for the following biomarkers of interest.
  * C-reactive protein (CRP)
  * -6 / Interleukin (IL) IL-8
  * Tumor necrosis factor-alpha (TNF-a)
Measuring stress with cancer | 6 weeks
  Stress will be measured using the Perceived Stress Scale (PSS). This 10-item measure is the most commonly used measure of perceptions of stress.
Measuring coping with cancer | 6 weeks
  Coping will be measured using the Cancer Behavior Inventory (CBI). The CBI is a 27-item measure of self-efficacy for coping with cancer.
Measuring affect with cancer | 6 weeks
  Affect will be measured using the Positive and Negative Affect Scale (PANAS). The PANAS is a 20 item scale measuring positive and negative affect.
Measuring emotional regulation with cancer | 6 weeks
  Emotion Regulation will be measured using the Emotion Regulation Questionnaire (ERQ). The ERQ is a 10-item self-report scale designed to measure use of strategies to alter emotion: reappraisal of cognitions and suppression of expressions.

CONTACTS AND LOCATIONS:
Overall Officials: Alia Crum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No